CLINICAL TRIAL: NCT06082869
Title: Evaluation and Comparison of a Novel Dentrifice Formulation on Plaque Removal
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Protegera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Protegera-2023-01
Record Dates: First submitted 2023-10-04; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: Randomized, single-center, examiner-blinded, parallel design clinical trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators performing plaque scoring, study coordinators entering plaque scores and handling data, and the statistician performing the data analysis were all blinded to the treatment regimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Protegera™ toothpaste (NaF), brushing twice daily for one minute
  Interventions: Drug: Protegera™ toothpaste (NaF)
- Control (Active Comparator): Crest™ Cavity Protection toothpaste (NaF), brushing twice daily for one minute
  Interventions: Drug: Crest™ Cavity Protection toothpaste (NaF)

INTERVENTIONS:
Drug: Protegera™ toothpaste (NaF) — Plaque Reduction
  Arms: Experimental
Drug: Crest™ Cavity Protection toothpaste (NaF) — Plaque Reduction
  Arms: Control

SUMMARY:
To evaluate and compare plaque removal efficacy and safety of a novel dentifrice formulation immediately after the first supervised use and following one week of twice, daily use at home.

DETAILED DESCRIPTION:
Study participants brushed their teeth for one minute, two times daily, for seven days.

Participants who met study entry criteria were randomized to either the test (Protegera™) or control (Crest™ Cavity Protection) toothpaste, and each were given the same straight, soft bristled toothbrush to use throughout the study.

On Day 1, participants were given an oral exam, and a pre-brushing plaque score was recorded. Participants then brushed their teeth for one minute under supervision, and a post-brushing plaque score was recorded.

On Day 7, participants were given an oral exam, and a pre-brushing plaque score was recorded. Participants then brushed their teeth for one minute under supervision, and a post-brushing plaque score was recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Have been males and females aged 18 to 69, in good general health.
2. Have read and signed an Informed Consent Form.
3. Have been in good health based on medical history review by the Principal Investigator.
4. Have had a minimum of 18 natural teeth with scorable facial and lingual surfaces. Teeth that were grossly carious, orthodontically banded, restorations such as crowns, veneers or implants, exhibit general cervical abrasion and/or enamel abrasion, or third molars were not included in the tooth count.
5. (If female of child bearing age) have been using an established method of birth control (systemic contraceptives such as birth control pills, injectable contraceptive or patch contraceptives, partner with vasectomy, condom with additional spermicide, IUD or abstinence).
6. Have had a mean full-mouth pre-brushing plaque score (Soparkar Modification1 of the Turesky Modification2 of the plaque index of Quigley and Hein.3) of ≥ 2.00 at the baseline visit.
7. Have agreed not to have a dental prophylaxis or any other elective, non-emergency dental procedures (other than those provided during the study) any time during the 7-day study.
8. Have been willing to refrain from all oral hygiene procedures (including chewing gum) for 24 hrs. and refrained from eating, drinking and smoking for approximately 2 hours prior to Visits 1 & 2.
9. Have agreed to refrain from use of all oral hygiene products (i.e., floss, mouthwash, etc.), other than the toothbrush and toothpaste supplied, for the duration of the 7-day study.
10. Have agreed to comply with the conditions and schedule of the study.

Exclusion Criteria:

1. Had any known allergies or sensitivities to marketed dentifrice or oral hygiene products.
2. Had any physical limitations or restrictions which might preclude normal tooth brushing.
3. Had existing serious medical condition or transmittable disease as determined after review of the medical history form. These will include but not be limited to: active hepatitis, tuberculosis, AIDS, asthma, bleeding disorder, diabetes, cirrhosis, leukemia, renal disease, sarcoidosis, vascular disease, thrush, or leukoplakia.
4. Self-reported as pregnant or nursing female.
5. Required antibiotic therapy within 30-days prior to study treatment.
6. Had a history of adverse effects, oral soft or hard tissue sensitivity, to any ingredient in the test materials.
7. Had received therapy with any medications, currently or within the last 30 days, which might interfere with the outcome of the study by affecting tissue condition, or salivation, particularly chronic therapy or long-term use, as determined by the investigator.
8. Had severe periodontal disease or being actively treated for periodontal disease.
9. Had fixed or removable orthodontic appliances, bridges, peri/oral piercings, or removable partial dentures.
10. Had significant oral soft tissue pathology based on a visual examination baseline.
11. Had evidence of poor oral hygiene or rampant dental caries or presence of extrinsic stain or calculus deposits that may interfere with plaque assessments.
12. Had received a dental prophylaxis within 30-days prior to Visit 1.
13. Had participated in another dental research study within 30-days prior to Visit 1.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Change In Dental Plaque | Day 1 and Day 7 of manual brushing
  Plaque measured on a scale of 0 to 5; 0 = No plaque; 5 = 2/3rd or more of tooth covered with plaque
Changes in oral soft or hard tissues | Day 1 and Day 7
  Examination of the oral cavity to determine any changes in color, soft tissue abrasion, texture or other irregularities

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L Milleman, DDS, MPA, Principal Investigator — Salus Research, Inc
Locations (1):
- Salus Research, Inc, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lobene RR, Soparkar PM, Newman MB. Use of dental floss. Effect on plaque and gingivitis. Clin Prev Dent. 1982 Jan-Feb;4(1):5-8. No abstract available. PMID 6980082
- [Result] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Result] QUIGLEY GA, HEIN JW. Comparative cleansing efficiency of manual and power brushing. J Am Dent Assoc. 1962 Jul;65:26-9. doi: 10.14219/jada.archive.1962.0184. No abstract available. PMID 14489483